CLINICAL TRIAL: NCT05942430
Title: Evaluation of the Effectiveness and Safety of Autologous Costal Osteochondral Transplantation in the Treatment of Talar Osteochondral Lesions: a Randomized Controlled Clinical Trial
Brief Title: Autologous Costal Osteochondral Transplantation for Talar Osteochondral Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Canjun Zeng, Director of the Department of Foot and Ankle Surgery, The Third Affiliated Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-Lunshen-017; YL202203 (Other Grant/Funding Number: The Dean's Fund)
Record Dates: First submitted 2023-06-18; First posted 2023-07-12 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Articular Cartilage Defect
Keywords: costa; autologous osteochondral transplantation; autologous osteoperiosteal transplantation; osteochondral lesion of the talus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The costa group (Experimental): Autologous costal osteochondral transplantation
  Interventions: Procedure: Autologous costal osteochondral transplantation
- The ilium group (Active Comparator): Autologous iliac osteoperiosteal transplantation
  Interventions: Procedure: Autologous iliac osteoperiosteal transplantation

INTERVENTIONS:
Procedure: Autologous costal osteochondral transplantation — Operating steps:
  1. Arthroscopic examination of the size and location of the talar osteochondral lesion;
  2. Make a transverse incision (approximately 4 cm long) at the osteochondral junction of the fifth or sixth rib, and harvest an osteochondral column from the rib;
  3. Thoroughly remove the talar osteochonral lesion through arthrotomy or Chevron osteotomy of the medial malleolus;
  4. Trim the autograft according to the size of the lesion;
  5. Fill the peri-lesion cavity with cancellous bone, and finally embed the costal osteochondral autograft into the talar defect, ensuring that the cartilage surface of the transplant to be flush with the normal talar cartilage around it;
  6. Suture the joint capsule or reduct and fix the medial malleolus, and close the incision layer by layer.
  Arms: The costa group
Procedure: Autologous iliac osteoperiosteal transplantation — Operating steps:
  1. Arthroscopic examination of the size and location of the talar osteochondral lesion;
  2. Make an incision along the anterior iliac crest. At the time of exposure, pay attention not to damage the periosteum. Obtain a cylindrical osteoperiosteal column by an appropriate-sized harvester tube.
  3. Thoroughly remove the talar osteochonral lesion through arthrotomy or Chevron osteotomy of the medial malleolus;
  4. Fill the peri-lesion cavity with cancellous bone, and finally embed the iliac osteoperiosteal autograft into the talar defect, ensuring that the periosteum surface of the transplant to be flush with the normal talar cartilage around it;
  5. Suture the joint capsule or reduct and fix the medial malleolus, and close the incision layer by layer.
  Arms: The ilium group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of autologous costal osteochondral transplantation in the treatment of Hepple Stage V talar osteochondral lesions, compared with autologous osteoperiosteal transplantation. The main question it aims to answer is:

• Whether autologous costal osteochondral transplantation can achieve better clinical outcomes and cartilage repair quality with lower donor site morbidity than autologous osteoperiosteal transplantation in the treatment of Hepple Stage V talar osteochondral lesions.

Participants will be randomly assigned to the intervention group (undergoing autologous costal osteochondral transplantation) or the control group (undergoing autologous osteoperiosteal transplantation). Both groups of participants will receive the same postoperative rehabilitation process and follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Hepple stage V talar osteochondral lesions with a lesion depth ≥5 mm and an AOFAS score ≤80 points;
* Failed conservative treatment for at least 6 months;
* Unilateral talar osteochondral lesions without corresponding lesions on the tibial side;
* Willingness to participate in this clinical trial and signing an informed consent form.

Exclusion Criteria:

* Combined with lower limb deformity.
* Combined with hip or knee joint diseases.
* Combined with ipsilateral ankle arthritis with joint space narrowing .
* Diagnosis of gouty arthritis of the ankle joint.
* Combined with osteoporosis (T score <-2.5).
* Other conditions considered inappropriate for participation in this clinical trial by the researchers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) ankle-hindfoot scale score | 24 months after surgery
  0-100

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) ankle-hindfoot scale score | 3, 6, 12 months after surgery
  0-100
International Cartilage Repair Society (ICRS) score | 12 months after surgery
  0-12; based on arthroscopic examination
Numeric Rating Scale (NRS) for ankle pain during walking | 3, 6, 12 and 24 months after surgery
  0-10
Foot and Ankle Ability Measure (FAAM) ADL subscale | 12 and 24 months after surgery
  0-100
Foot and Ankle Ability Measure (FAAM) Sports subscale | 12 and 24 months after surgery
  0-100
Tegner score | 12 and 24 months after surgery
  0-10
Patients' satisfaction degree | 24 months after surgery
  0-10
Bone union | 3 months after surgery or later
  Based on computed tomography scan
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score | 12 and 24 months after surgery
  0-100; based on magnetic resonance imaging
Numeric Rating Scale (NRS) for donor-site pain | 1, 2, 3, 6, 12 and 24 months after surgery
  0-10
Any other complications | 1, 2, 3, 6, 12 and 24 months after surgery
  Any other complications

CONTACTS AND LOCATIONS:
Overall Officials: Canjun Zeng, PhD, Principal Investigator — The Third Affiliated Hospital of Southern Medical University
Locations (1):
- The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No